CLINICAL TRIAL: NCT03480711
Title: Modified Trabeculectomy With an Extended Subscleral Tunnel Versus Conventional Trabeculectomy for Management of Primary Open Angle Glaucoma (POAG)
Brief Title: Modified Trabeculectomy With an ESST Versus Conventional SST for Management of Primary Open Angle Glaucoma
Acronym: POAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab mahmoud abdelhamid mohamed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Rehab mahmoud abdelhamid mohamed, assistant lecturer of ophthalmology,ophthalmology department, medical school, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-38-2018
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Primary Open-angle Glaucoma
Keywords: subscleral trabeculectomy; extended subscleral tunnel; mitomycinC
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Population Groups; Trabeculectomy

STUDY DESIGN:
Intervention Model Description: Randomized non-controlled comparative prospective interventional study
Who Masked: Participant, Outcomes Assessor
Masking Description: participants are going to be randomly assigned into two groups outcomes assessor will asses
  1. visual acuity and BCVA
  2. IOP using Goldmann applanation tonometry
  3. slit-lamp and fundus examination of cup-disc ratio,
  4. Ultrasound Biomicroscopy (UBM) to assese ostium patency and extent of bleb area will be done once after 6 weeks post-operatively.
  5. Colored photography of the filtering blebs will be performed for grading. Bleb grading will be classified according moorfields grading scale
  6. Perimetry will be performed at the end of follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): 20 eyes of 20 patients of uncontrolled POAG administrated intervention will be subscleral trabeculectomy (SST) single surgeon, using retrobulbar anaesthesia with 2% lidocaine, will be performed in all surgeries. Following insertion of a lid speculum, a 10/0 silk bridle suture is inserted at superior limbus if required. In group (A) a conjunctival incision is made at the limbus to create a fornix-based conjunctival flap. A half thickness scleral flap (4 × 4 mm) are created and dissected into the clear cornea. A cellulose microsponge soaked in 0.3 mg/ml MMC solution (Mitomycin-C) is applied to the under surface of the scleral flap over a wide posterior area for 2 ml
  Interventions: Procedure: SST in group (A)
- group (B) (Experimental): 20 eyes of 20 patients of uncontrolled POAG d Administrated intervention will be ESST another longitudinal scleral groove will be created in the center of the deep scleral bed area measured about 1.5 × 6 mm.In both groups, standard trabeculectomy of equal size (two bites aside) is created by a Kelly punch ( 1 mm)
  Interventions: Procedure: trabeculectomy with ESST in group (B)

INTERVENTIONS:
Procedure: SST in group (A) — group (A) single surgeon, using retrobulbar anaesthesia with 2% lidocaine, will be performed in all surgeries. Following insertion of a lid speculum, a 10/0 silk bridle suture is inserted at superior limbus if required. In group (A) a conjunctival incision is made at the limbus to create a fornix-based conjunctival flap. A half thickness scleral flap (4 × 4 mm) are created and dissected into the clear cornea. A cellulose microsponge soaked in 0.3 mg/ml MMC solution (Mitomycin-C) is applied to the under surface of the scleral flap over a wide posterior area for 2 ml
  Other Names: subscleral trabeculectomy; conventional trabeculectomy
  Arms: Group (A)
Procedure: trabeculectomy with ESST in group (B) — group (B), another longitudinal scleral groove will be created in the center of the deep scleral bed area measured about 1.5 × 6 mm.In both groups, standard trabeculectomy of equal size (two bites aside) is created by a Kelly punch ( 1 mm)
  Other Names: modified trabeculectomy; extended subscleral tunnel
  Arms: group (B)

SUMMARY:
* To evaluate prospectively the surgical outcome in terms of intraocular pressure control, potential advantages, disadvantages, success rate, complications and bleb morphology of this modified trabeculectomy with an extended subscleral tunnel (ESST) in comparison to the conventional subscleral trabeculectomy (SST) in management of uncontrolled primary open angle glaucoma.
* This study will recruit 40 eyes of (40) candidate patients with primary open angle glaucoma (POAG) who are indicated for surgery.
* The candidate patients will be recruited into 2 equal comparative groups. In group (A) 20 eyes (20 patients) who will undergo conventional (SST) with intraoperative mitomycin C (MMC) (0.03%) and group (B); 20 eyes of 20 patients will undergo trabeculectomy with an ESST also with intraoperative adjunctive MMC (0.03%).

DETAILED DESCRIPTION:
* Different surgical procedures were developed and the principle behind them was to establish a fistula between the anterior chamber and the subconjunctival space to permit the aqueous humour to exit the eye.
* Subscleral trabeculectomy has remained the most commonly performed glaucoma surgery to which the newer operations are compared.Although this procedure is very effective in reducing intraocular pressure (IOP) immediately, surgical failure has often been observed over time due to fibrosis of the surgical site and resultant non-filtering bleb. -Improvement of the complication profile and the efficacy of glaucoma filtering surgery is still a major concern for glaucoma surgeons.Therefore, several modifications, combinations, and new techniques of subscleral trabeculectomy have been described.
* In the current study, a fornix-based conjunctival flap will be fashioned in an attempt to encourage more posterior drainage. In this modified trabeculectomy technique, an additional small perpendicular strip of sclera is removed extending from the AC to 2 mm beyond the edge of the scleral flap thus creating an extended subscleral trabeculectomy facilitating aqueous passage into the posterior subconjunctival space.

ELIGIBILITY:
Inclusion Criteria:

* Patients with POAG aged from (40- 70) years who are candidate for glaucoma surgery with BCVA ≥ 3/60 to be able to perform visual field testing.
* Non- compliant patients to the medical treatment willing for follow-up visits for at least 6 months post-operatively .

Exclusion Criteria:

* Congenital, traumatic, neovascular, uveitic glaucomas or cases with angle closure glaucoma (ACG) associated with shallow AC.
* Undergoing simultaneous cataract surgery.
* Previous vitreo-retinal surgery including vitrectomy and buckling surgery.
* Other pre-existing ocular cicatrizing diseases.
* Corneal abnormality that precluded reliable applanation tonometry.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
change from baseline intraocular pressure at first day postoperative | day one postoperatively
  mmHg
change from baseline intraocular pressure at 4 weeks | , 4 weeks.
  mmHg
change from baseline intraocular pressure at 6 weeks Ultrasound bimicroscopy (UBM) | 6 weeks post-operatively.
  mm Hg
change from baseline intraocular pressure at 3 months | 3 months postoperatively
  mmHg
change from baseline intraocular pressure at 6 months | 6 months postoperatively
  mmHg

SECONDARY OUTCOMES:
change from baseline best corrected visual acuity (BCVA) at 6 months | at the end of 6 months
  logarithm of minimal angle of resolution (log MAR)
extent of filtering bleb area by ultrasound of bio-microscopy (UBM) | 6 weeks postoperatively
  width, depth and height of filtering bleb area in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Riham S Allam, MD, FRCS GL, Principal Investigator — Associate Professor of Ophthalmology , Cairo university; Karim A Raafat, MD, Principal Investigator — Professor of Ophthalmology , Cairo university; Rehab M Mohamed, MD, Principal Investigator — lecturer of Ophthalmology , Cairo university
Locations (1):
- Faculty of medicind, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study protocol Statistical analysis plan within 6 months after completing the study

REFERENCES:
- [Background] El Sayyad F, Belmekki M, Helal M, Khalil M, El-Hamzawey H, Hisham M. Simultaneous subconjunctival and subscleral mitomycin-C application in trabeculectomy. Ophthalmology. 2000 Feb;107(2):298-301; discussion 302. doi: 10.1016/s0161-6420(99)00097-4. PMID 10690829
- [Background] Nuijts RM, Vernimmen RC, Webers CA. Mitomycin C primary trabeculectomy in primary glaucoma of white patients. J Glaucoma. 1997 Oct;6(5):293-7. PMID 9327347